CLINICAL TRIAL: NCT02872142
Title: Pilot Study to Evaluate the Efficacy and Safety of Plasma Exchange With Albutein® 5% in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Efficacy and Safety of Plasma Exchange With Albutein® 5% in Participants With Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBI1501
Record Dates: First submitted 2016-08-11; First posted 2016-08-19 (Estimated); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Albumins; Solutions; Perfusion; Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Albutein 5% (Experimental): Plasma exchanges (PEs) with albutein 5% as a replacement solution during an intensive treatment phase of two PEs per week over 3 weeks followed by maintenance treatment phase of weekly PE for 21 weeks. The dose of albutein 5% for replacement following plasma removal was calculated based on gender, weight, and the hematocrit of the participant.
  Interventions: Biological: Albutein 5%; Procedure: Plasma Exchange

INTERVENTIONS:
Biological: Albutein 5% — Albutein is manufactured from human plasma. The dose of Albutein 5% for replacement following plasma removal will be calculated based on gender, weight, and the hematocrit of the participant.
  Other Names: Albutein 5% solution for perfusion
Procedure: Plasma Exchange — Plasma Exchange will be performed using albutein 5% as the replacement solution.

SUMMARY:
This is a pilot, phase 2, prospective, open-label, single-arm study to evaluate disease progression, forced vital capacity, and the safety and tolerability of plasma exchange (PE) using Albutein® 5% in participants with amyotrophic lateral sclerosis (ALS).

DETAILED DESCRIPTION:
This is a phase 2, prospective, open-label, single-arm pilot study to evaluate the efficacy and safety of PE with Albutein® 5% in participants with ALS. The planned enrollment is 10 participants who have a definite, possible, or probable diagnosis of ALS, according to the revised El Escorial criteria. Enrolled participants will be treated with PE using Albutein 5% as a replacement solution during an Intensive Treatment Phase (2 PEs per week over 3 weeks) followed by a Maintenance Treatment Phase (weekly PE for 21 weeks) for a total treatment duration of 6 months. A 6-month follow up will begin after the last PE.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Subjects over 18 years of age and less than 70 years old
* Subjects with a possible, probable-lab supported, probable, or definite diagnosis of Amyotrophic Lateral Sclerosis (ALS), according to the revised El Escorial criteria
* Subjects having experienced their first ALS symptoms within 18 months prior to recruitment/consent
* Forced Vital Capacity > 70%
* Subjects must be medically suitable for study participation and willing to comply with all planned aspects of the protocol, including blood sampling, at the time of inclusion in the study.

Exclusion Criteria:

* Subjects with pre-existing clinically significant lung disease not attributable to ALS
* Subjects diagnosed with other neurodegenerative diseases or diseases associated with other motor neuron dysfunction
* Participation in another investigational product study within one month prior to screening
* Females who are pregnant, breastfeeding, or, if of child-bearing potential, unwilling to practice a highly effective method of contraception (oral, injectable or implanted hormonal methods of contraception, placement of an intrauterine device or intrauterine system, condom or occlusive cap with spermicidal foam/ gel/ film/ cream/ suppository, male sterilization, or true abstinence) throughout the study
* Difficult or problematic peripheral vein access and inability to implant a central catheter which would make continuous Plasma exchange (PE) not feasible as per the visit protocol
* Contraindication to undergo PE or subject has abnormal coagulation parameters at the discretion of the Outpatient Apheresis Unit team, including but not limited to:

  1. Thrombocytopenia (platelets <100,000/ microliter [μL])
  2. Fibrinogen <1.5 gram per liter (g/L)
  3. International Normalized Ratio >1.5
  4. Beta-blocker treatment and bradycardia <50 beats/min
  5. Treatment with angiotensin-converting enzyme inhibitors which may increase the risk of allergic reactions, unless a preventive change in hypotensive treatment occurs prior to enrollment
* History of anaphylaxis or severe systemic response to any plasma-derived albumin preparation, component of Albutein® 5%, or other blood product(s)
* Subjects unable to interrupt treatment with acetylsalicylic acid, other oral antiplatelet, or anticoagulant
* Renal dysfunction by elevated creatinine concentration >2 milligram per deciliter (mg/dL)
* Presence of heart disease that contraindicates PE treatment, including ischemic cardiopathy and congestive heart failure
* Presence of prior behavioural disorders requiring pharmacological intervention with less than 3 months of stable treatment
* Mentally challenged subject who cannot give independent informed consent
* Any condition that would complicate compliance with the study protocol (i.e., illness with the expectation of less than one year survival, abuse of drugs or alcohol, etc.)

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at a single study center in the Unites States from 29 August 2016 to 15 August 2019.
Pre-assignment Details: Participants with diagnosis of amyotrophic lateral sclerosis (ALS) were enrolled to receive plasma exchanges with albutein 5% as a replacement solution as per the protocol defined schedule for 24 weeks.
Period: Overall Study
Arm/Group | Albutein 5%
Started | 12
Completed | 6
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Participant Decision | 3

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any amount of the study drug.
Groups:
- Albutein 5%: PEs with albutein 5% as a replacement solution during an intensive treatment phase of two PEs per week over 3 weeks followed by maintenance treatment phase of weekly PE for 21 weeks. The dose of albutein 5% for replacement following plasma removal was calculated based on gender, weight, and the hematocrit of the participant.
Arm/Group | Albutein 5%
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.98 (7.590)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) Score
Description: The ALSFRS-R includes 12 questions to assess the self-sufficiency of participants in 3 sub-domains: bulbar function (questions 1-3), fine and gross motor function (questions 4-9), and respiratory function (question 10-12). Aspects of nourishment, personal care, personal autonomy, and communication were also evaluated. Each task was graded on a five-point scale from 0 (incapable) to 4 (normal ability), with total score range from 0 (worst) to 48 (best). A positive change from Baseline indicates improvement.
Time Frame: Baseline (Week 0), Weeks 4, 12, 25, 36, and 48
Population: Evaluable Population included all participants who received at least one PE treatment with albutein 5% and also had at least one baseline determination and a measurement of a primary efficacy variable at a subsequent visit. Number analyzed is the number of participants with data available for analyses at the given time point.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Albutein 5%
Number analyzed (Participants) | 12
units on scale
  Baseline | 39.8 (5.88)
  Change at Week 4 | -1.3 (3.17)
  Change at Week 12: number analyzed (Participants) | 11
  Change at Week 12 | -2.5 (1.97)
  Change at Week 25: number analyzed (Participants) | 7
  Change at Week 25 | -5.0 (5.03)
  Change at Week 36: number analyzed (Participants) | 8
  Change at Week 36 | -9.3 (6.39)
  Change at Week 48: number analyzed (Participants) | 7
  Change at Week 48 | -8.9 (4.74)

2. Primary Outcome: Change From Baseline in Percent Predicted Forced Vital Capacity (FVC)
Description: The FVC measured the volume of air that can forcibly be exhaled through a spirometer after a full inspiration. It was expressed in a percentage of actual FVC over the expected FVC result in the general population, calculated as: Percent predicted FVC (in %) = [(observed FVC in liters)/(predicted FVC in liters)]*100.
Time Frame: Baseline (Week 0), Weeks 4, 12, 25, 36, and 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of predicted FVC
Arm/Group | Albutein 5%
Number analyzed (Participants) | 12
percentage of predicted FVC
  Baseline | 89.7 (16.26)
  Change at Week 4 | -2.6 (4.78)
  Change at Week 12: number analyzed (Participants) | 11
  Change at Week 12 | -6.3 (5.50)
  Change at Week 25: number analyzed (Participants) | 7
  Change at Week 25 | -13.9 (7.01)
  Change at Week 36: number analyzed (Participants) | 8
  Change at Week 36 | -19.4 (12.44)
  Change at Week 48: number analyzed (Participants) | 7
  Change at Week 48 | -21.0 (14.83)

3. Secondary Outcome: Change From Baseline in Cognitive Function as Assessed by Behaviour Status Sub-scale Score of the Amyotrophic Lateral Sclerosis - Cognitive Behavioural Screen (ALS-CBS) Test
Description: ALS-CBS test is composed of two sections: the cognitive screening section and behavioural changes section. The section of behavioural changes consists of behaviour status and symptom status sub-scales. Behaviour status sub-scale consists of a questionnaire with 15 items assessed by the caretaker. Each item was scored on a scale ranging from 0 (worst) to 3 (best) yielding a total 0= large changes to 45= no changes. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Week 0), Weeks 25, and 48
Population: Evaluable Population included all participants who received at least one PE treatment with albutein 5% and also had at least one baseline determination and measurement of a primary efficacy variable at a subsequent visit. Number analyzed is the number of participants with data available for analyses at the given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Albutein 5%
Number analyzed (Participants) | 11
units on a scale
  Baseline | 41.7 (3.44)
  Change at Week 25: number analyzed (Participants) | 6
  Change at Week 25 | -1.8 (2.79)
  Change at Week 48: number analyzed (Participants) | 6
  Change at Week 48 | -8.5 (5.28)

4. Secondary Outcome: Change From Baseline in Cognitive Function as Assessed by Symptom Status Sub-scale Score of the Amyotrophic Lateral Sclerosis - Cognitive Behavioral Screen (ALS-CBS) Test
Description: ALS-CBS test is composed of two sections: cognitive screening section and behavioural changes section. The section of behavioural changes consists of behaviour status and symptom status sub-scales. Cognitive function assessed by symptom status sub-scale is reported, which consists of 4 additional questions related to current behavioural symptoms (depression, anxiety, fatigue, and emotional liability). Each question was scored as 0= the presence of symptoms and 1= no current symptoms, giving a total subscale score between 0 and 4. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Week 0), Weeks 25, and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Albutein 5%
Number analyzed (Participants) | 11
units on scale
  Baseline | 3.5 (0.69)
  Change at Week 25: number analyzed (Participants) | 6
  Change at Week 25 | -0.2 (0.75)
  Change at Week 48: number analyzed (Participants) | 6
  Change at Week 48 | -0.2 (1.33)

5. Secondary Outcome: Change From Baseline in Cognitive Function as Assessed by Cognitive Screening Section Score of the Amyotrophic Lateral Sclerosis - Cognitive Behavioral Screen (ALS-CBS) Test
Description: ALS-CBS test is composed of two sections: cognitive screening section and behavioural changes section. Cognitive function is evaluated using cognitive screening section which consists of: attention (complex orders, mental sums, language, and eye movement); concentration (inversion of numeric series); follow-up and monitoring (reverse sequences, alphabet, number and letter sequencing); and initiation and recovery (nomination). The individual items were scored from 0-5, and the total score ranges from 0-20, where 0= cognitive impairment, 20= no apparent cognitive impairment. A positive change from baseline indicates improvement.
Time Frame: Baseline (Week 0), Weeks 25, and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Albutein 5%
Number analyzed (Participants) | 11
units on scale
  Baseline | 16.4 (5.12)
  Change at Week 25: number analyzed (Participants) | 6
  Change at Week 25 | 1.0 (2.76)
  Change at Week 48: number analyzed (Participants) | 6
  Change at Week 48 | 0.8 (2.79)

6. Secondary Outcome: Change From Baseline in the Motor Evoked Potential in Thenar and Hypothenar Eminence and Anterior Tibialis Muscle Determined by Electromyography (EMG)
Description: Surface EMG was performed to record motor evoked potential in the distal muscles of the upper limbs (thenar and hypothenar eminence) and dorsiflexor muscles of the lower limbs (anterior tibialis) after electrical stimulation on the median, ulnar, and external popliteal sciatic nerve. The data for motor evoked potential (in millivolt [mv]) is reported for thenar muscles of both upper limbs and hypothenar muscle of the upper right limb and anterior tibialis of the both lower limbs.
Time Frame: Baseline (Week 0), Weeks 4, 12, 25, 36, and 48
Population: Evaluable Population included all participants who received at least one PE treatment with albutein 5% and also had at least one baseline determination and a measurement of a primary efficacy variable at a subsequent visit. Number analyzed is the number of participants with data available for the specific category at the given time point.
Measure: Mean (Standard Deviation); unit: millivolt (mV)
Arm/Group | Albutein 5%
Number analyzed (Participants) | 12
millivolt (mV)
  Right Tibialis Anterior, Baseline | 4.1 (2.36)
  Right Tibialis Anterior, Change at Week 4: number analyzed (Participants) | 11
  Right Tibialis Anterior, Change at Week 4 | -0.4 (1.49)
  Right Tibialis Anterior, Change at Week 12: number analyzed (Participants) | 11
  Right Tibialis Anterior, Change at Week 12 | -0.1 (1.85)
  Right Tibialis Anterior, Change at Week 25: number analyzed (Participants) | 7
  Right Tibialis Anterior, Change at Week 25 | -1.3 (3.19)
  Right Tibialis Anterior, Change at Week 36: number analyzed (Participants) | 6
  Right Tibialis Anterior, Change at Week 36 | -0.7 (3.72)
  Right Tibialis Anterior, Change at Week 48: number analyzed (Participants) | 6
  Right Tibialis Anterior, Change at Week 48 | -1.6 (3.46)
  Left Tibialis Anterior, Baseline | 4.2 (2.02)
  Left Tibialis Anterior, Change at Week 4 | -0.7 (1.72)
  Left Tibialis Anterior, Change at Week 12: number analyzed (Participants) | 11
  Left Tibialis Anterior, Change at Week 12 | -0.6 (2.13)
  Left Tibialis Anterior, Change at Week 25: number analyzed (Participants) | 7
  Left Tibialis Anterior, Change at Week 25 | -0.7 (2.69)
  Left Tibialis Anterior, Change at Week 36: number analyzed (Participants) | 6
  Left Tibialis Anterior, Change at Week 36 | -0.8 (3.58)
  Left Tibialis Anterior, Change at Week 48: number analyzed (Participants) | 6
  Left Tibialis Anterior, Change at Week 48 | -1.3 (3.36)
  Right Thenar Eminence, Baseline | 4.3 (3.01)
  Right Thenar Eminence, Change at Week4: number analyzed (Participants) | 10
  Right Thenar Eminence, Change at Week4 | -0.3 (1.18)
  Right Thenar Eminence, Change at Week 12: number analyzed (Participants) | 9
  Right Thenar Eminence, Change at Week 12 | -0.6 (1.29)
  Right Thenar Eminence, Change at Week 25: number analyzed (Participants) | 6
  Right Thenar Eminence, Change at Week 25 | -1.3 (2.39)
  Right Thenar Eminence, Change at Week 36: number analyzed (Participants) | 5
  Right Thenar Eminence, Change at Week 36 | -1.5 (2.40)
  Right Thenar Eminence, Change at Week 48: number analyzed (Participants) | 6
  Right Thenar Eminence, Change at Week 48 | -2.1 (2.78)
  Left Thenar Eminence, Baseline: number analyzed (Participants) | 10
  Left Thenar Eminence, Baseline | 3.8 (3.20)
  Left Thenar Eminence, Change at Week 4: number analyzed (Participants) | 9
  Left Thenar Eminence, Change at Week 4 | 0.2 (1.63)
  Left Thenar Eminence, Change at Week 12: number analyzed (Participants) | 8
  Left Thenar Eminence, Change at Week 12 | -0.2 (1.34)
  Left Thenar Eminence, Change at Week 25: number analyzed (Participants) | 6
  Left Thenar Eminence, Change at Week 25 | 0.3 (2.61)
  Left Thenar Eminence, Change at Week 36: number analyzed (Participants) | 4
  Left Thenar Eminence, Change at Week 36 | -1.4 (2.48)
  Left Thenar Eminence, Change at Week 48: number analyzed (Participants) | 3
  Left Thenar Eminence, Change at Week 48 | -0.9 (1.83)
  Right Hypothenar Eminence, Baseline: number analyzed (Participants) | 11
  Right Hypothenar Eminence, Baseline | 6.4 (2.50)
  Right Hypothenar Eminence, Change at Week 4: number analyzed (Participants) | 11
  Right Hypothenar Eminence, Change at Week 4 | -0.5 (1.23)
  Right Hypothenar Eminence, Change at Week 12: number analyzed (Participants) | 10
  Right Hypothenar Eminence, Change at Week 12 | -1.1 (0.82)
  Right Hypothenar Eminence, Change at Week 25: number analyzed (Participants) | 7
  Right Hypothenar Eminence, Change at Week 25 | -1.9 (2.24)
  Right Hypothenar Eminence, Change at Week 36: number analyzed (Participants) | 6
  Right Hypothenar Eminence, Change at Week 36 | -2.6 (2.29)
  Right Hypothenar Eminence, Change at Week 48: number analyzed (Participants) | 5
  Right Hypothenar Eminence, Change at Week 48 | -3.2 (1.41)

7. Secondary Outcome: Evaluation of Quality of Life Using the Amyotrophic Lateral Sclerosis Assessment Questionnaire 40 (ALSA-Q40) Test Dimension Score
Description: The ALS questionnaire consists of 40 items grouped into 5 representative dimensions associated with quality of life. The first four dimensions were: physical mobility (questions 1-10), activities of daily living (questions 11- 20), food and drink (questions 21-23), communication (questions 24-30) and emotional function (questions 31-40), refer to deficits and subsequent disabilities as a result of the disease. The fifth scale (emotional functioning) reflects how the participant is facing his/her physical deterioration emotionally. Each item is scored from 0 to 4 according to a gradation of symptom onset frequency (never, rarely, sometimes, often, always). From raw scores, an index from 0 to 100 is obtained for each dimension, which make comparisons with the other dimensions possible as well as a straightforward interpretation of the results (0 = better state of health as measured by the questionnaire;100 = poorer state of health). A negative change from Baseline indicates improvement.
Time Frame: Weeks 25 and 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Albutein 5%
Number analyzed (Participants) | 12
units on a scale
  Physical mobility Week 25: number analyzed (Participants) | 7
  Physical mobility Week 25 | 23.6 (17.61)
  Physical mobility Week 48: number analyzed (Participants) | 7
  Physical mobility Week 48 | 20.7 (15.26)
  ADL/independence Week 25: number analyzed (Participants) | 7
  ADL/independence Week 25 | 25.4 (15.91)
  ADL/independence Week 48: number analyzed (Participants) | 7
  ADL/independence Week 48 | 27.9 (14.82)
  Eating and drinking Week 25: number analyzed (Participants) | 7
  Eating and drinking Week 25 | 8.3 (21.52)
  Eating and drinking Week 48: number analyzed (Participants) | 7
  Eating and drinking Week 48 | 14.3 (29.94)
  Communication Week 25: number analyzed (Participants) | 7
  Communication Week 25 | 7.7 (11.92)
  Communication Week 48: number analyzed (Participants) | 7
  Communication Week 48 | 9.7 (12.49)
  Emotional functioning Week 25: number analyzed (Participants) | 7
  Emotional functioning Week 25 | 8.9 (14.50)
  Emotional functioning Week 48: number analyzed (Participants) | 7
  Emotional functioning Week 48 | 11.4 (17.13)

8. Secondary Outcome: Change From Baseline in Plasma Human Apolipoprotein Levels
Description: The levels of human Apolipoprotein (ApoE) in plasma were measured by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline (Week 0), before and after PE procedure at Weeks 4, 12, 24, and before PE for Weeks 36 and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Albutein 5%
Number analyzed (Participants) | 12
nanogram per milliliter (ng/mL)
  Baseline | 6753.8 (3549.07)
  Before PE, Change at Week 4 | 645.9 (2122.00)
  After PE, Change at Week 4 | -3978.2 (2749.25)
  Before PE, Change at Week 12: number analyzed (Participants) | 10
  Before PE, Change at Week 12 | 611.5 (3014.69)
  After PE, Change at Week 12: number analyzed (Participants) | 10
  After PE, Change at Week 12 | -3504.2 (3434.69)
  Before PE, Change at Week 24: number analyzed (Participants) | 7
  Before PE, Change at Week 24 | -555.3 (2782.05)
  After PE, Change at Week 24: number analyzed (Participants) | 7
  After PE, Change at Week 24 | -4711.3 (3142.53)
  Before PE, Change at Week 36: number analyzed (Participants) | 8
  Before PE, Change at Week 36 | 643.0 (2306.95)
  Before PE, Change at Week 48: number analyzed (Participants) | 6
  Before PE, Change at Week 48 | 861.0 (4242.19)

9. Secondary Outcome: Change From Baseline in Plasma Cytokine Panel Levels
Description: The plasma cytokine panel includes: transforming growth factor (TGF) beta1, TGF beta2, TGF beta3, interferon (IFN) gamma, interleukins (IL)-1beta, IL-1Ra, IL-6, IL-8, IL-10, IL-12 p70, IL-17A, IFN-γ-inducible protein (IP)-10, human monocyte chemoattractant protein (MCP)-1, macrophage-derived chemokine (MDC), macrophage inflammatory protein (MIP)-1-alpha, MIP-1-beta, tumor necrosis factor (TNF)-alpha, soluble cluster of differentiation (CD) 40 ligand (sCD40L), fractalkine. The level of each of these cytokines are reported as categories. Only categories with values above the level of detection are reported.
Time Frame: Baseline (Week 0), before and after PE procedure at Weeks 4, 12, 24, and before PE for Weeks 36 and 48
Population: Evaluable Population included all participants who received at least one PE treatment with albutein 5% and also had at least one baseline determination and measurement of a primary efficacy variable at a subsequent visit. Number analyzed is the number of participants with detectable values for the analyses of the specific category at the given time point.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Albutein 5%
Number analyzed (Participants) | 12
picogram per milliliter (pg/mL)
  TGF beta1; Baseline | 9998.9 (5811.61)
  TGF beta1; Before PE, Change at Week 4 | -1302.4 (7269.45)
  TGF beta1; After PE, Change at Week 4 | -5922.8 (5490.19)
  TGF beta1; Before PE, Change at Week 12: number analyzed (Participants) | 10
  TGF beta1; Before PE, Change at Week 12 | 1238.6 (7838.89)
  TGF beta1; After PE, Change at Week 12: number analyzed (Participants) | 10
  TGF beta1; After PE, Change at Week 12 | -5476.7 (5453.16)
  TGF beta1; Before PE, Change at Week 24: number analyzed (Participants) | 7
  TGF beta1; Before PE, Change at Week 24 | -86.6 (5270.57)
  TGF beta1; After PE, Change at Week 24: number analyzed (Participants) | 7
  TGF beta1; After PE, Change at Week 24 | -4966.4 (4711.24)
  TGF beta1; Before PE, Change at Week 36: number analyzed (Participants) | 8
  TGF beta1; Before PE, Change at Week 36 | -1698.5 (6124.07)
  TGF beta1; Before PE, Change at Week 48: number analyzed (Participants) | 6
  TGF beta1; Before PE, Change at Week 48 | -1160.5 (5942.4)
  TGF beta2; Baseline | 465.8 (247.85)
  TGF beta2; Before PE, Change at Week 4 | -22.1 (323.20)
  TGF beta2; After PE, Change at Week 4 | -244.4 (228.25)
  TGF beta2; Before PE, Change at Week 12: number analyzed (Participants) | 10
  TGF beta2; Before PE, Change at Week 12 | 64.4 (329.48)
  TGF beta2; After PE, Change at Week 12: number analyzed (Participants) | 10
  TGF beta2; After PE, Change at Week 12 | -207.9 (203.96)
  TGF beta2; Before PE, Change at Week 24: number analyzed (Participants) | 7
  TGF beta2; Before PE, Change at Week 24 | 5.8 (259.18)
  TGF beta2; After PE, Change at Week 24: number analyzed (Participants) | 6
  TGF beta2; After PE, Change at Week 24 | -220.4 (236.01)
  TGF beta2; Before PE, Change at Week 36: number analyzed (Participants) | 8
  TGF beta2; Before PE, Change at Week 36 | -62.5 (270.98)
  TGF beta2; Before PE, Change at Week 48: number analyzed (Participants) | 6
  TGF beta2; Before PE, Change at Week 48 | -28.1 (262.15)
  TGF beta3; Baseline: number analyzed (Participants) | 3
  TGF beta3; Baseline | 63.70 (0.000)
  IFN gamma; Baseline: number analyzed (Participants) | 5
  IFN gamma; Baseline | 16.22 (9.024)
  IFN gamma; Before PE, Change at Week 4: number analyzed (Participants) | 1
  IFN gamma; Before PE, Change at Week 4 | 8.80 (NA) — Standard deviation (SD) was not estimable as there was only one participant.
  IFN gamma; Before PE, Change at Week 12: number analyzed (Participants) | 2
  IFN gamma; Before PE, Change at Week 12 | -5.70 (15.415)
  IFN gamma; Before PE, Change at Week 24: number analyzed (Participants) | 2
  IFN gamma; Before PE, Change at Week 24 | -4.70 (6.647)
  IFN gamma; Before PE, Change at Week 36: number analyzed (Participants) | 2
  IFN gamma; Before PE, Change at Week 36 | 8.40 (3.677)
  IFN gamma; Before PE, Change at Week 48: number analyzed (Participants) | 1
  IFN gamma; Before PE, Change at Week 48 | 9.60 (NA) — SD was not estimable as there was only one participant.
  Interleukin (IL)-1beta; Baseline: number analyzed (Participants) | 1
  Interleukin (IL)-1beta; Baseline | 16.10 (NA) — SD was not estimable as there was only one participant.
  IL-1Ra; Baseline | 56.7 (44.19)
  IL-1Ra; Before PE, Change at Week 4: number analyzed (Participants) | 10
  IL-1Ra; Before PE, Change at Week 4 | -7.4 (33.93)
  IL-1Ra; After PE, Change at Week 4: number analyzed (Participants) | 11
  IL-1Ra; After PE, Change at Week 4 | -17.5 (17.70)
  IL-1Ra; Before PE, Change at Week 12: number analyzed (Participants) | 9
  IL-1Ra; Before PE, Change at Week 12 | 1.1 (31.99)
  IL-1Ra; After PE, Change at Week 12: number analyzed (Participants) | 9
  IL-1Ra; After PE, Change at Week 12 | -5.7 (24.09)
  IL-1Ra; Before PE, Change at Week 24: number analyzed (Participants) | 6
  IL-1Ra; Before PE, Change at Week 24 | 3.3 (13.36)
  IL-1Ra; After PE, Change at Week 24: number analyzed (Participants) | 5
  IL-1Ra; After PE, Change at Week 24 | 1.2 (13.79)
  IL-1Ra; Before PE, Change at Week 36: number analyzed (Participants) | 8
  IL-1Ra; Before PE, Change at Week 36 | 0.5 (10.31)
  IL-1Ra; Before PE, Change at Week 48: number analyzed (Participants) | 6
  IL-1Ra; Before PE, Change at Week 48 | 3.6 (8.79)
  IL-6; Baseline: number analyzed (Participants) | 6
  IL-6; Baseline | 160.7 (132.82)
  IL-6; Before PE, Change at Week 4: number analyzed (Participants) | 4
  IL-6; Before PE, Change at Week 4 | -0.9 (128.32)
  IL-6; After PE, Change at Week 4: number analyzed (Participants) | 3
  IL-6; After PE, Change at Week 4 | -112.3 (64.94)
  IL-6; Before PE, Change at Week 12: number analyzed (Participants) | 4
  IL-6; Before PE, Change at Week 12 | 6.5 (121.65)
  IL-6; After PE, Change at Week 12: number analyzed (Participants) | 2
  IL-6; After PE, Change at Week 12 | -78.7 (130.04)
  IL-6; Before PE, Change at Week 24: number analyzed (Participants) | 2
  IL-6; Before PE, Change at Week 24 | -43.0 (23.26)
  IL-6; After PE, Change at Week 24: number analyzed (Participants) | 1
  IL-6; After PE, Change at Week 24 | -166.9 (NA) — SD was not estimable as there was only one participant.
  IL-6; Before PE, Change at Week 36: number analyzed (Participants) | 3
  IL-6; Before PE, Change at Week 36 | -18.8 (39.89)
  IL-6; Before PE, Change at Week 48: number analyzed (Participants) | 2
  IL-6; Before PE, Change at Week 48 | 3.3 (16.55)
  IL-8; Baseline: number analyzed (Participants) | 7
  IL-8; Baseline | 48.4 (57.66)
  IL-8; Before PE, Change at Week 4: number analyzed (Participants) | 4
  IL-8; Before PE, Change at Week 4 | -4.2 (32.27)
  IL-8; After PE, Change at Week 4: number analyzed (Participants) | 4
  IL-8; After PE, Change at Week 4 | -45.5 (24.99)
  IL-8; Before PE, Change at Week 12: number analyzed (Participants) | 4
  IL-8; Before PE, Change at Week 12 | 3.9 (39.30)
  IL-8; After PE, Change at Week 12: number analyzed (Participants) | 3
  IL-8; After PE, Change at Week 12 | -38.4 (9.98)
  IL-8; Before PE, Change at Week 24: number analyzed (Participants) | 3
  IL-8; Before PE, Change at Week 24 | -9.3 (7.64)
  IL-8; After PE, Change at Week 24: number analyzed (Participants) | 2
  IL-8; After PE, Change at Week 24 | -24.8 (35.00)
  IL-8; Before PE, Change at Week 36: number analyzed (Participants) | 3
  IL-8; Before PE, Change at Week 36 | -8.3 (10.10)
  IL-8; Before PE, Change at Week 48: number analyzed (Participants) | 3
  IL-8; Before PE, Change at Week 48 | -1.2 (4.41)
  IL-10; Baseline: number analyzed (Participants) | 9
  IL-10; Baseline | 10.34 (13.056)
  IL-10; Before PE, Change at Week 4: number analyzed (Participants) | 4
  IL-10; Before PE, Change at Week 4 | -4.70 (9.731)
  IL-10; After PE, Change at Week 4: number analyzed (Participants) | 5
  IL-10; After PE, Change at Week 4 | -4.46 (12.398)
  IL-10; Before PE, Change at Week 12: number analyzed (Participants) | 6
  IL-10; Before PE, Change at Week 12 | -0.25 (2.638)
  IL-10; After PE, Change at Week 12: number analyzed (Participants) | 4
  IL-10; After PE, Change at Week 12 | -0.45 (2.626)
  IL-10; Before PE, Change at Week 24: number analyzed (Participants) | 4
  IL-10; Before PE, Change at Week 24 | -0.50 (1.354)
  IL-10; After PE, Change at Week 24: number analyzed (Participants) | 4
  IL-10; After PE, Change at Week 24 | -1.13 (1.181)
  IL-10; Before PE, Change at Week 36: number analyzed (Participants) | 4
  IL-10; Before PE, Change at Week 36 | 1.38 (2.720)
  IL-10; Before PE, Change at Week 48: number analyzed (Participants) | 2
  IL-10; Before PE, Change at Week 48 | 2.50 (0.707)
  IL-12 p70; Baseline: number analyzed (Participants) | 6
  IL-12 p70; Baseline | 11.95 (2.026)
  IL-12 p70; Before PE, Change at Week 12: number analyzed (Participants) | 1
  IL-12 p70; Before PE, Change at Week 12 | 2.10 (NA) — SD was not estimable as there was only one participant.
  IL-12 p70; Before PE, Change at Week 24: number analyzed (Participants) | 2
  IL-12 p70; Before PE, Change at Week 24 | -1.25 (3.041)
  IL-12 p70; After PE, Change at Week 24: number analyzed (Participants) | 2
  IL-12 p70; After PE, Change at Week 24 | -2.15 (1.768)
  IL-12 p70; Before PE, Change at Week 36: number analyzed (Participants) | 2
  IL-12 p70; Before PE, Change at Week 36 | 0.90 (1.273)
  IL-12 p70; Before PE, Change at Week 48: number analyzed (Participants) | 2
  IL-12 p70; Before PE, Change at Week 48 | 2.15 (4.313)
  IL-17A; Baseline: number analyzed (Participants) | 6
  IL-17A; Baseline | 5.28 (4.351)
  IL-17A; Before PE, Change at Week 4: number analyzed (Participants) | 2
  IL-17A; Before PE, Change at Week 4 | -1.90 (1.556)
  IL-17A; After PE, Change at Week 4: number analyzed (Participants) | 4
  IL-17A; After PE, Change at Week 4 | 2.48 (1.132)
  IL-17A; Before PE, Change at Week 12: number analyzed (Participants) | 1
  IL-17A; Before PE, Change at Week 12 | 1.90 (NA) — SD was not estimable as there was only one participant.
  IL-17A; After PE, Change at Week 12: number analyzed (Participants) | 2
  IL-17A; After PE, Change at Week 12 | 2.35 (0.636)
  IL-17A; Before PE, Change at Week 24: number analyzed (Participants) | 2
  IL-17A; Before PE, Change at Week 24 | -0.40 (0.000)
  IL-17A; After PE, Change at Week 24: number analyzed (Participants) | 3
  IL-17A; After PE, Change at Week 24 | 1.33 (1.617)
  IL-17A; Before PE, Change at Week 36: number analyzed (Participants) | 2
  IL-17A; Before PE, Change at Week 36 | 1.30 (0.283)
  IL-17A; Before PE, Change at Week 48: number analyzed (Participants) | 1
  IL-17A; Before PE, Change at Week 48 | 3.00 (NA) — SD was not estimable as there was only one participant.
  IP-10; Baseline | 407.0 (133.95)
  IP-10; Before PE, Change at Week 4 | -38.4 (104.78)
  IP-10; After PE, Change at Week 4 | 27.9 (153.91)
  IP-10; Before PE, Change at Week 12: number analyzed (Participants) | 10
  IP-10; Before PE, Change at Week 12 | -7.7 (122.81)
  IP-10; After PE, Change at Week 12: number analyzed (Participants) | 10
  IP-10; After PE, Change at Week 12 | -2.7 (144.21)
  IP-10; Before PE, Change at Week 24: number analyzed (Participants) | 7
  IP-10; Before PE, Change at Week 24 | -2.1 (152.60)
  IP-10; After PE, Change at Week 24: number analyzed (Participants) | 7
  IP-10; After PE, Change at Week 24 | -42.7 (166.87)
  IP-10; Before PE, Change at Week 36: number analyzed (Participants) | 8
  IP-10; Before PE, Change at Week 36 | 25.6 (129.09)
  IP-10; Before PE, Change at Week 48: number analyzed (Participants) | 6
  IP-10; Before PE, Change at Week 48 | -23.8 (156.50)
  Human Monocyte Chemoattractant Protein-1 (MCP-1); Baseline | 239.1 (69.94)
  MCP-1; Before PE, Change at Week 4 | 44.5 (81.02)
  MCP-1; After PE, Change at Week 4 | 102.2 (117.01)
  MCP-1; Before PE, Change at Week 12: number analyzed (Participants) | 10
  MCP-1; Before PE, Change at Week 12 | 51.6 (118.85)
  MCP-1; After PE, Change at Week 12: number analyzed (Participants) | 10
  MCP-1; After PE, Change at Week 12 | 73.7 (113.07)
  MCP-1; Before PE, Change at Week 24: number analyzed (Participants) | 7
  MCP-1; Before PE, Change at Week 24 | 63.2 (130.31)
  MCP-1; After PE, Change at Week 24: number analyzed (Participants) | 7
  MCP-1; After PE, Change at Week 24 | 40.1 (33.36)
  MCP-1; Before PE, Change at Week 36: number analyzed (Participants) | 8
  MCP-1; Before PE, Change at Week 36 | -41.3 (64.66)
  MCP-1; Before PE, Change at Week 48: number analyzed (Participants) | 6
  MCP-1; Before PE, Change at Week 48 | -25.8 (37.85)
  Macrophage-Derived Chemokine (MDC); Baseline | 547.7 (178.98)
  MDC; Before PE, Change at Week 4 | 57.6 (135.92)
  MDC; After PE, Change at Week 4 | 20.7 (220.90)
  MDC; Before PE, Change at Week 12: number analyzed (Participants) | 10
  MDC; Before PE, Change at Week 12 | 41.8 (133.82)
  MDC; After PE, Change at Week 12: number analyzed (Participants) | 10
  MDC; After PE, Change at Week 12 | -4.2 (164.87)
  MDC; Before PE, Change at Week 24: number analyzed (Participants) | 7
  MDC; Before PE, Change at Week 24 | 98.5 (134.08)
  MDC; After PE, Change at Week 24: number analyzed (Participants) | 7
  MDC; After PE, Change at Week 24 | -73.1 (182.85)
  MDC; Before PE, Change at Week 36: number analyzed (Participants) | 8
  MDC; Before PE, Change at Week 36 | 41.4 (139.68)
  MDC; Before PE, Change at Week 48: number analyzed (Participants) | 6
  MDC; Before PE, Change at Week 48 | -16.3 (121.81)
  Macrophage Inflammatory Protein (MIP-1) alpha; Baseline: number analyzed (Participants) | 7
  Macrophage Inflammatory Protein (MIP-1) alpha; Baseline | 7.54 (4.109)
  MIP-1 alpha; Before PE, Change at Week 4: number analyzed (Participants) | 4
  MIP-1 alpha; Before PE, Change at Week 4 | -0.43 (4.971)
  MIP-1 alpha; After PE, Change at Week 4: number analyzed (Participants) | 3
  MIP-1 alpha; After PE, Change at Week 4 | -2.50 (4.590)
  MIP-1 alpha; Before PE, Change at Week 12: number analyzed (Participants) | 5
  MIP-1 alpha; Before PE, Change at Week 12 | 0.46 (3.580)
  MIP-1 alpha; After PE, Change at Week 12: number analyzed (Participants) | 3
  MIP-1 alpha; After PE, Change at Week 12 | -1.10 (2.691)
  MIP-1 alpha; Before PE, Change at Week 24: number analyzed (Participants) | 2
  MIP-1 alpha; Before PE, Change at Week 24 | -0.80 (0.283)
  MIP-1 alpha; After PE, Change at Week 24: number analyzed (Participants) | 1
  MIP-1 alpha; After PE, Change at Week 24 | -1.50 (NA) — SD was not estimable as there was only one participant.
  MIP-1 alpha; Before PE, Change at Week 36: number analyzed (Participants) | 3
  MIP-1 alpha; Before PE, Change at Week 36 | 0.63 (0.351)
  MIP-1 alpha; Before PE, Change at Week 48: number analyzed (Participants) | 2
  MIP-1 alpha; Before PE, Change at Week 48 | 1.05 (0.636)
  MIP-1 beta; Baseline | 60.33 (24.913)
  MIP-1 beta; Before PE, Change at Week 4 | -1.17 (18.954)
  MIP-1 beta; After PE, Change at Week 4 | 3.97 (33.788)
  MIP-1 beta; Before PE, Change at Week 12: number analyzed (Participants) | 10
  MIP-1 beta; Before PE, Change at Week 12 | -1.48 (15.869)
  MIP-1 beta; After PE, Change at Week 12: number analyzed (Participants) | 10
  MIP-1 beta; After PE, Change at Week 12 | 3.33 (31.079)
  MIP-1 beta; Before PE, Change at Week 24: number analyzed (Participants) | 7
  MIP-1 beta; Before PE, Change at Week 24 | -3.97 (13.444)
  MIP-1 beta; After PE, Change at Week 24: number analyzed (Participants) | 7
  MIP-1 beta; After PE, Change at Week 24 | -8.61 (17.402)
  MIP-1 beta; Before PE, Change at Week 36: number analyzed (Participants) | 8
  MIP-1 beta; Before PE, Change at Week 36 | 0.33 (16.394)
  MIP-1 beta; Before PE, Change at Week 48: number analyzed (Participants) | 6
  MIP-1 beta; Before PE, Change at Week 48 | -6.58 (12.213)
  Tumor Necrosis Factor-Alpha (TNF alpha); Baseline: number analyzed (Participants) | 9
  Tumor Necrosis Factor-Alpha (TNF alpha); Baseline | 16.80 (4.832)
  TNF alpha; Before PE, Change at Week 4: number analyzed (Participants) | 9
  TNF alpha; Before PE, Change at Week 4 | -1.38 (5.803)
  TNF alpha; After PE, Change at Week 4: number analyzed (Participants) | 9
  TNF alpha; After PE, Change at Week 4 | 1.11 (5.766)
  TNF alpha; Before PE, Change at Week 12: number analyzed (Participants) | 7
  TNF alpha; Before PE, Change at Week 12 | -0.06 (6.450)
  TNF alpha; After PE, Change at Week 12: number analyzed (Participants) | 7
  TNF alpha; After PE, Change at Week 12 | -0.07 (3.645)
  TNF alpha; Before PE, Change at Week 24: number analyzed (Participants) | 4
  TNF alpha; Before PE, Change at Week 24 | -2.77 (2.229)
  TNF alpha; After PE, Change at Week 24: number analyzed (Participants) | 4
  TNF alpha; After PE, Change at Week 24 | 0.03 (3.673)
  TNF alpha; Before PE, Change at Week 36: number analyzed (Participants) | 5
  TNF alpha; Before PE, Change at Week 36 | -0.74 (3.970)
  TNF alpha; Before PE, Change at Week 48: number analyzed (Participants) | 3
  TNF alpha; Before PE, Change at Week 48 | -2.37 (4.474)
  sCD40L; Baseline | 137.3 (83.74)
  sCD40L; Before PE, Change at Week 4 | 31.6 (160.97)
  sCD40L; After PE, Change at Week 4: number analyzed (Participants) | 11
  sCD40L; After PE, Change at Week 4 | -52.3 (81.20)
  sCD40L; Before PE, Change at Week 12: number analyzed (Participants) | 10
  sCD40L; Before PE, Change at Week 12 | 48.9 (138.73)
  sCD40L; After PE, Change at Week 12: number analyzed (Participants) | 9
  sCD40L; After PE, Change at Week 12 | -31.2 (91.56)
  sCD40L; Before PE, Change at Week 24: number analyzed (Participants) | 7
  sCD40L; Before PE, Change at Week 24 | 47.8 (188.88)
  sCD40L; After PE, Change at Week 24: number analyzed (Participants) | 7
  sCD40L; After PE, Change at Week 24 | -49.8 (56.50)
  sCD40L; Before PE, Change at Week 36: number analyzed (Participants) | 8
  sCD40L; Before PE, Change at Week 36 | -2.4 (39.84)
  sCD40L; Before PE, Change at Week 48: number analyzed (Participants) | 6
  sCD40L; Before PE, Change at Week 48 | -30.1 (93.64)
  Fractalkine; Baseline: number analyzed (Participants) | 9
  Fractalkine; Baseline | 240.6 (69.12)
  Fractalkine; Before PE, Change at Week 4: number analyzed (Participants) | 6
  Fractalkine; Before PE, Change at Week 4 | -63.6 (111.89)
  Fractalkine; After PE, Change at Week 4: number analyzed (Participants) | 3
  Fractalkine; After PE, Change at Week 4 | -32.1 (73.32)
  Fractalkine; Before PE, Change at Week 12: number analyzed (Participants) | 6
  Fractalkine; Before PE, Change at Week 12 | 2.0 (103.06)
  Fractalkine; After PE, Change at Week 12: number analyzed (Participants) | 1
  Fractalkine; After PE, Change at Week 12 | -35.0 (NA) — SD was not estimable as there was only one participant.
  Fractalkine; Before PE, Change at Week 24: number analyzed (Participants) | 4
  Fractalkine; Before PE, Change at Week 24 | -10.5 (34.89)
  Fractalkine; After PE, Change at Week 24: number analyzed (Participants) | 2
  Fractalkine; After PE, Change at Week 24 | -43.3 (5.59)
  Fractalkine; Before PE, Change at Week 36: number analyzed (Participants) | 3
  Fractalkine; Before PE, Change at Week 36 | -5.7 (81.28)
  Fractalkine; Before PE, Change at Week 48: number analyzed (Participants) | 3
  Fractalkine; Before PE, Change at Week 48 | 15.0 (104.63)

10. Secondary Outcome: Change From Baseline in Cerebrospinal Fluid (CSF) Human Apolipoprotein Levels
Description: The levels of human Apolipoprotein (ApoE) in CSF were measured by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline (Week 0), Weeks 12, and 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Albutein 5%
Number analyzed (Participants) | 12
ng/mL
  Baseline | 3877.7 (1479.73)
  Change at Week 12: number analyzed (Participants) | 11
  Change at Week 12 | -188.0 (889.06)
  Change at Week 25: number analyzed (Participants) | 7
  Change at Week 25 | 20.0 (743.95)

11. Secondary Outcome: Change From Baseline in CSF Cytokine Panel Levels
Description: The CSF cytokine panel includes: TGF beta1, TGF beta2, TGF beta3, IFN gamma, IL-1beta, IL-1Ra, IL-6, IL-8, IL-10, IL-12 p70, IL-17A, IP-10, MCP-1, MDC, MIP-1 alpha, MIP-1 beta, TNF alpha, sCD40L, fractalkine. The level of each of these cytokines are reported as categories. Only categories with values above the level of detection are reported.
Time Frame: Baseline (Week 0), Weeks 12, and 25
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albutein 5%
Number analyzed (Participants) | 12
pg/mL
  TGF beta2; Baseline | 224.73 (36.830)
  TGF beta2; Change at Week 12: number analyzed (Participants) | 11
  TGF beta2; Change at Week 12 | -8.38 (27.358)
  TGF beta2; Change at Week 25: number analyzed (Participants) | 7
  TGF beta2; Change at Week 25 | 4.24 (26.517)
  IL-1Ra; Baseline: number analyzed (Participants) | 1
  IL-1Ra; Baseline | 11.20 (NA) — SD was not estimable as there was only one participant.
  IL-8; Baseline | 28.71 (6.575)
  IL-8; Change at Week 12: number analyzed (Participants) | 11
  IL-8; Change at Week 12 | -0.30 (4.323)
  IL-8; Change at Week 25: number analyzed (Participants) | 7
  IL-8; Change at Week 25 | 2.11 (5.498)
  IL-12 p70; Baseline: number analyzed (Participants) | 1
  IL-12 p70; Baseline | 3.80 (NA) — SD was not estimable as there was only one participant.
  IL-17A; Baseline | 20.16 (4.870)
  IL-17A; Change at Week 12: number analyzed (Participants) | 11
  IL-17A; Change at Week 12 | -0.84 (3.211)
  IL-17A; Change at Week 25: number analyzed (Participants) | 7
  IL-17A; Change at Week 25 | -2.61 (5.591)
  IP-10; Baseline | 493.6 (239.39)
  IP-10; Change at Week 12: number analyzed (Participants) | 11
  IP-10; Change at Week 12 | -38.4 (99.46)
  IP-10; Change at Week 25: number analyzed (Participants) | 7
  IP-10; Change at Week 25 | -30.6 (218.26)
  MCP-1; Baseline | 1325.7 (331.09)
  MCP-1; Change at Week 12: number analyzed (Participants) | 11
  MCP-1; Change at Week 12 | -80.6 (169.01)
  MCP-1; Change at Week 25: number analyzed (Participants) | 7
  MCP-1; Change at Week 25 | 30.5 (235.17)
  MDC; Baseline: number analyzed (Participants) | 2
  MDC; Baseline | 9.70 (2.970)
  MDC; Change at Week 12: number analyzed (Participants) | 1
  MDC; Change at Week 12 | 0.00 (NA) — SD was not estimable as there was only one participant.
  MIP-1 beta; Baseline | 13.95 (4.555)
  MIP-1 beta; Change at Week 12: number analyzed (Participants) | 11
  MIP-1 beta; Change at Week 12 | 0.18 (3.393)
  MIP-1 beta; Change at Week 25: number analyzed (Participants) | 7
  MIP-1 beta; Change at Week 25 | -0.44 (3.054)
  TNF alpha; Baseline: number analyzed (Participants) | 8
  TNF alpha; Baseline | 3.83 (1.809)
  TNF alpha; Change at Week 12: number analyzed (Participants) | 6
  TNF alpha; Change at Week 12 | 0.40 (1.717)
  TNF alpha; Change at Week 25: number analyzed (Participants) | 4
  TNF alpha; Change at Week 25 | -0.85 (1.731)
  sCD40L; Baseline: number analyzed (Participants) | 4
  sCD40L; Baseline | 4.13 (2.955)
  sCD40L; Change at Week 12: number analyzed (Participants) | 1
  sCD40L; Change at Week 12 | -5.50 (NA) — SD was not estimable as there was only one participant.
  sCD40L; Change at Week 25: number analyzed (Participants) | 1
  sCD40L; Change at Week 25 | 1.80 (NA) — SD was not estimable as there was only one participant.
  Fractalkine; Baseline: number analyzed (Participants) | 3
  Fractalkine; Baseline | 16.17 (8.776)
  Fractalkine; Change at Week 12: number analyzed (Participants) | 2
  Fractalkine; Change at Week 12 | 0.00 (0.000)
  Fractalkine; Change at Week 25: number analyzed (Participants) | 2
  Fractalkine; Change at Week 25 | 0.00 (0.000)

12. Secondary Outcome: Change From Baseline in Plasma Beta-methylamino-L-alanine (BMAA) Levels
Description: Plasma BMAA levels at baseline and over the course of treatment at each evaluation visit were measured to identify reductions in BMAA levels, which could potentially be correlated with disease progression or a halt in disease progression. Analysis was performed using a Thermo TSQ Quantiva triple-stage quadrupole mass spectrometer.
Time Frame: Baseline (Week 0), before and after PE procedure at Weeks 4, 12, 24, and before PE for Weeks 36 and 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Albutein 5%
Number analyzed (Participants) | 12
ng/mL
  Baseline | NA (NA) — Data is not available as BMAA concentration levels were below the level of detection.
  Change at Week 4: number analyzed (Participants) | 11
  Change at Week 4 | NA (NA) — Data is not available as BMAA concentration levels were below the level of detection.
  Change at Week 12: number analyzed (Participants) | 11
  Change at Week 12 | NA (NA) — Data is not available as BMAA concentration levels were below the level of detection.
  Change at Week 24: number analyzed (Participants) | 11
  Change at Week 24 | NA (NA) — Data is not available as BMAA concentration levels were below the level of detection.
  Change at Week 25: number analyzed (Participants) | 7
  Change at Week 25 | NA (NA) — Data is not available as BMAA concentration levels were below the level of detection.
  Change at Week 48: number analyzed (Participants) | 6
  Change at Week 48 | NA (NA) — Data is not available as BMAA concentration levels were below the level of detection.

13. Secondary Outcome: Change From Cerebrospinal Fluid (CSF) Beta-methylamino-L-alanine (BMAA) Levels
Description: CSF BMAA levels at baseline and over the course of treatment at each evaluation visit were measured to identify reductions in BMAA levels, which could potentially be correlated with disease progression or a halt in disease progression. Analysis was performed using a Thermo TSQ Quantiva triple quadrupole mass spectrometer.
Time Frame: Baseline (Week 0), Weeks 12, and 25
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Albutein 5%
Number analyzed (Participants) | 12
ng/mL
  Baseline | NA (NA) — Data is not available as BMAA concentration levels were below the level of detection.
  Change at Week 12: number analyzed (Participants) | 11
  Change at Week 12 | NA (NA) — Data is not available as BMAA concentration levels were below the level of detection.
  Change at Week 25: number analyzed (Participants) | 7
  Change at Week 25 | NA (NA) — Data is not available as BMAA concentration levels were below the level of detection.

14. Secondary Outcome: Change From Baseline in Absolute Leukocyte Count
Description: The immune population profile in ALS participants was assessed by flow cytometry following whole blood staining by Western Blot (WB) for the absolute leukocyte count. Absolute leukocyte count (10^3 cells/microliter) was analyzed for neutrophils, lymphocytes, CD14+ monocytes, CD3+CD4+ T cells, CD3+CD8+ T cells, CD19+ B cells and CD56+ natural killer (NK) cells.
Time Frame: Baseline, Weeks 4, 12, and 48
Population: Evaluable Population included all participants who received at least one PE treatment with albutein 5% and also had at least one baseline determination and a measurement of a primary efficacy variable at a subsequent visit. Number analyzed is the number of participants with data available for analyses of the specific category at the given time point.
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliter
Arm/Group | Albutein 5%
Number analyzed (Participants) | 12
10^3 cells/microliter
  Absolute leukocyte count neutrophils, Baseline | 4.18 (1.359)
  Absolute leukocyte count neutrophils, Change at Week 4 | -0.42 (0.828)
  Absolute leukocyte count neutrophils, Change at Week 12: number analyzed (Participants) | 11
  Absolute leukocyte count neutrophils, Change at Week 12 | 0.47 (0.732)
  Absolute leukocyte count neutrophils, Change at Week 48: number analyzed (Participants) | 6
  Absolute leukocyte count neutrophils, Change at Week 48 | 0.08 (1.731)
  Absolute leukocyte count lymphocytes, Baseline | 2.08 (0.881)
  Absolute leukocyte count lymphocytes, Change at Week 4 | 0.41 (0.703)
  Absolute leukocyte count lymphocytes, Change at Week 12: number analyzed (Participants) | 11
  Absolute leukocyte count lymphocytes, Change at Week 12 | 0.38 (1.158)
  Absolute leukocyte count lymphocytes, Change at Week 48: number analyzed (Participants) | 6
  Absolute leukocyte count lymphocytes, Change at Week 48 | 0.95 (0.914)
  Absolute leukocyte count CD14+ monocytes, Baseline | 0.49 (0.188)
  Absolute leukocyte count CD14+ monocytes, Change at Week 4 | -0.05 (0.157)
  Absolute leukocyte count CD14+ monocytes, Change at Week 12: number analyzed (Participants) | 11
  Absolute leukocyte count CD14+ monocytes, Change at Week 12 | 0.07 (0.228)
  Absolute leukocyte count CD14+ monocytes, Change at Week 48: number analyzed (Participants) | 6
  Absolute leukocyte count CD14+ monocytes, Change at Week 48 | 0.03 (0.225)
  Absolute leukocyte count CD3+CD4+ T cells, Baseline | 1.01 (0.403)
  Absolute leukocyte count CD3+CD4+ T cells, Change at Week 4 | 0.19 (0.390)
  Absolute leukocyte count CD3+CD4+ T cells, Change at Week12: number analyzed (Participants) | 11
  Absolute leukocyte count CD3+CD4+ T cells, Change at Week12 | 0.27 (0.666)
  Absolute leukocyte count CD3+CD4+ T cells, Change at Week 48: number analyzed (Participants) | 6
  Absolute leukocyte count CD3+CD4+ T cells, Change at Week 48 | 0.43 (0.641)
  Absolute leukocyte count CD3+CD8+ T cells, Baseline | 0.38 (0.266)
  Absolute leukocyte count CD3+CD8+ T cells, Change at Week 4 | 0.01 (0.144)
  Absolute leukocyte count CD3+CD8+ T cells, Change at Week 12: number analyzed (Participants) | 11
  Absolute leukocyte count CD3+CD8+ T cells, Change at Week 12 | 0.05 (0.242)
  Absolute leukocyte count CD3+CD8+ T cells, Change at Week 48: number analyzed (Participants) | 6
  Absolute leukocyte count CD3+CD8+ T cells, Change at Week 48 | 0.13 (0.186)
  Absolute leukocyte count CD19+ B cells, Baseline | 0.07 (0.089)
  Absolute leukocyte count CD19+ B cells, Change at Week 4 | 0.00 (0.043)
  Absolute leukocyte count CD19+ B cells, Change at Week 12: number analyzed (Participants) | 11
  Absolute leukocyte count CD19+ B cells, Change at Week 12 | 0.03 (0.110)
  Absolute leukocyte count CD19+ B cells, Change at Week 48: number analyzed (Participants) | 6
  Absolute leukocyte count CD19+ B cells, Change at Week 48 | 0.00 (0.063)
  Absolute leukocyte count CD56+ NK cells, Baseline | 0.22 (0.127)
  Absolute leukocyte count CD56+ NK cells Change at Week 4 | 0.05 (0.124)
  Absolute leukocyte count CD56+ NK cells, Change at Week 12: number analyzed (Participants) | 11
  Absolute leukocyte count CD56+ NK cells, Change at Week 12 | 0.03 (0.101)
  Absolute leukocyte count CD56+ NK cells, Change at Week 48: number analyzed (Participants) | 6
  Absolute leukocyte count CD56+ NK cells, Change at Week 48 | 0.07 (0.103)

15. Secondary Outcome: Change From Baseline in Immune Population Profile
Description: The immune population profile includes: Leukocyte panel (neutrophils, lymphocytes, CD14+ monos, CD3+CD4+ T cells, CD3+CD8+ T cells, CD19+ B cells, CD56+ NK cells). Regulatory T cells (Treg panel) (CD4+FoxP3+CD127low/, CD4+FoxP3+CD127low/-CD39+, CD4+FoxP3+CD127low/-CD45RA, CD4+FoxP3+CD127low/-CD152+), Myeloid-Derived Suppressor Cells (MDSC) (panel: CD14+CD15- monocytic MDSCs, CD14+CD15- monocytic MDSCs, CD124+ monocytic MDSCs, CD14-CD15+ granulocytic MDSCs, CD124+ granulocytic MDSCs, CD14-CD15- immature MDSCs, CD124+ immature MDSCs), Monocyte panel (CD14+CD16+, CD14+human leukocyte antigen-D related (HLA-DR)+ CD11b, CD14+HLA-DR+ CD163+, CD14+HLA-DR+ CX3CR1+). Data for each of these were reported as categories. Only categories with values above the level of detection are reported.
Time Frame: Baseline, Weeks 4, 12, and 48
Population: Evaluable Population included all participants who received at least one PE treatment with albutein 5% and also had at least one baseline determination and a measurement of a primary efficacy variable at a subsequent visit. Number analyzed is the number of participants with detectable values for analyses of the specific category at the given time point.
Measure: Mean (Standard Deviation); unit: percentage of CD45+ cells
Arm/Group | Albutein 5%
Number analyzed (Participants) | 12
percentage of CD45+ cells
  Leukocyte panel: neutrophils; Baseline | 68.13 (11.672)
  Leukocyte panel: neutrophils; Change at Week 4 | -6.58 (9.457)
  Leukocyte panel: neutrophils; Change at Week 12: number analyzed (Participants) | 11
  Leukocyte panel: neutrophils; Change at Week 12 | -0.26 (12.391)
  Leukocyte panel: neutrophils; Change at Week 48: number analyzed (Participants) | 6
  Leukocyte panel: neutrophils; Change at Week 48 | -10.08 (13.188)
  Leukocyte panel: lymphocytes; Baseline | 23.48 (11.681)
  Leukocyte panel: lymphocytes; Change at Week 4 | 7.12 (10.026)
  Leukocyte panel: lymphocytes; Change at Week 12: number analyzed (Participants) | 11
  Leukocyte panel: lymphocytes; Change at Week 12 | 1.17 (10.531)
  Leukocyte panel: lymphocytes; Change at Week 48: number analyzed (Participants) | 6
  Leukocyte panel: lymphocytes; Change at Week 48 | 11.94 (15.553)
  Leukocyte panel: CD14+ monos; Baseline | 6.49 (1.832)
  Leukocyte panel: CD14+ monos; Change at Week 4 | -0.92 (2.592)
  Leukocyte panel: CD14+ monos; Change at Week 12: number analyzed (Participants) | 11
  Leukocyte panel: CD14+ monos; Change at Week 12 | -0.31 (2.329)
  Leukocyte panel: CD14+ monos; Change at Week 48: number analyzed (Participants) | 6
  Leukocyte panel: CD14+ monos; Change at Week 48 | 0.34 (3.424)
  Leukocyte panel: CD3+CD4+ T cells; Baseline | 11.58 (6.274)
  Leukocyte panel: CD3+CD4+ T cells; Change at Week 4 | 4.77 (5.956)
  Leukocyte panel: CD3+CD4+ T cells; Change at Week 12: number analyzed (Participants) | 11
  Leukocyte panel: CD3+CD4+ T cells; Change at Week 12 | 0.17 (7.230)
  Leukocyte panel: CD3+CD4+ T cells; Change at Week 48: number analyzed (Participants) | 6
  Leukocyte panel: CD3+CD4+ T cells; Change at Week 48 | 5.46 (10.954)
  Leukocyte panel: CD3+CD8+ T cells; Baseline | 3.71 (2.473)
  Leukocyte panel: CD3+CD8+ T cells; Change at Week 4 | 1.12 (1.529)
  Leukocyte panel: CD3+CD8+ T cells; Change at Week 12: number analyzed (Participants) | 11
  Leukocyte panel: CD3+CD8+ T cells; Change at Week 12 | 0.14 (1.303)
  Leukocyte panel: CD3+CD8+ T cells; Change at Week 48: number analyzed (Participants) | 6
  Leukocyte panel: CD3+CD8+ T cells; Change at Week 48 | 1.64 (3.179)
  Leukocyte panel: CD19+ B cells; Baseline | 2.12 (1.312)
  Leukocyte panel: CD19+ B cells; Change at Week 4 | 1.06 (1.420)
  Leukocyte panel: CD19+ B cells; Change at Week 12: number analyzed (Participants) | 11
  Leukocyte panel: CD19+ B cells; Change at Week 12 | 0.56 (1.240)
  Leukocyte panel: CD19+ B cells; Change at Week 48: number analyzed (Participants) | 6
  Leukocyte panel: CD19+ B cells; Change at Week 48 | 1.88 (1.931)
  Leukocyte panel: CD56+ NK cells; Baseline | 3.80 (2.610)
  Leukocyte panel: CD56+ NK cells; Change at Week 4 | -0.04 (1.417)
  Leukocyte panel: CD56+ NK cells; Change at Week 12: number analyzed (Participants) | 11
  Leukocyte panel: CD56+ NK cells; Change at Week 12 | -0.17 (2.051)
  Leukocyte panel: CD56+ NK cells; Change at Week 48: number analyzed (Participants) | 6
  Leukocyte panel: CD56+ NK cells; Change at Week 48 | 0.92 (4.419)
  Regulatory T cells (Treg panel): CD4+FoxP3+CD127low/-; Baseline | 0.5717 (0.40475)
  Treg panel: CD4+FoxP3+CD127low/-; Change at Week 4 | -0.0267 (0.21641)
  Treg panel: CD4+FoxP3+CD127low/-; Change at Week 12: number analyzed (Participants) | 11
  Treg panel: CD4+FoxP3+CD127low/-; Change at Week 12 | -0.1648 (0.41184)
  Treg panel: CD4+FoxP3+CD127low/-; Change at Week 48: number analyzed (Participants) | 6
  Treg panel: CD4+FoxP3+CD127low/-; Change at Week 48 | -0.0658 (0.35043)
  Treg panel: CD4+FoxP3+CD127low/-CD39+; Baseline: number analyzed (Participants) | 7
  Treg panel: CD4+FoxP3+CD127low/-CD39+; Baseline | 0.1196 (0.08932)
  Treg panel: CD4+FoxP3+CD127low/-CD39+; Change at Week 4: number analyzed (Participants) | 2
  Treg panel: CD4+FoxP3+CD127low/-CD39+; Change at Week 4 | 0.1845 (0.10536)
  Treg panel: CD4+FoxP3+CD127low/-CD39+; Change at Week 12: number analyzed (Participants) | 1
  Treg panel: CD4+FoxP3+CD127low/-CD39+; Change at Week 12 | -0.1300 (NA) — SD was not estimable as there was only one participant.
  Treg panel: CD4+FoxP3+CD127low/-CD39+; Change at Week 48: number analyzed (Participants) | 2
  Treg panel: CD4+FoxP3+CD127low/-CD39+; Change at Week 48 | -0.0850 (0.25314)
  Treg panel: CD4+FoxP3+CD127low/-CD45RA; Baseline | 0.4953 (0.34120)
  Treg panel: CD4+FoxP3+CD127low/-CD45RA; Change at Week 4 | 0.6278 (2.17115)
  Treg panel: CD4+FoxP3+CD127low/-CD45RA; Change at Week 12: number analyzed (Participants) | 11
  Treg panel: CD4+FoxP3+CD127low/-CD45RA; Change at Week 12 | -0.1296 (0.34452)
  Treg panel: CD4+FoxP3+CD127low/-CD45RA; Change at Week 48: number analyzed (Participants) | 6
  Treg panel: CD4+FoxP3+CD127low/-CD45RA; Change at Week 48 | -0.0420 (0.29646)
  Treg panel: CD4+FoxP3+CD127low/-CD152+; Baseline: number analyzed (Participants) | 11
  Treg panel: CD4+FoxP3+CD127low/-CD152+; Baseline | 0.2028 (0.17937)
  Treg panel: CD4+FoxP3+CD127low/-CD152+; Change at Week 4: number analyzed (Participants) | 11
  Treg panel: CD4+FoxP3+CD127low/-CD152+; Change at Week 4 | -0.0282 (0.10316)
  Treg panel: CD4+FoxP3+CD127low/-CD152+; Change at Week 12: number analyzed (Participants) | 8
  Treg panel: CD4+FoxP3+CD127low/-CD152+; Change at Week 12 | -0.1100 (0.16162)
  Treg panel: CD4+FoxP3+CD127low/-CD152+; Change at Week 48: number analyzed (Participants) | 5
  Treg panel: CD4+FoxP3+CD127low/-CD152+; Change at Week 48 | 0.0490 (0.32648)
  Myeloid-Derived Suppressor Cells (MDSC) panel: CD14+CD15- monocytic MDSCs; Baseline | 0.3207 (0.25371)
  Myeloid-Derived Suppressor Cells (MDSC) panel: CD14+CD15- monocytic MDSCs; Change at Week 4: number analyzed (Participants) | 10
  Myeloid-Derived Suppressor Cells (MDSC) panel: CD14+CD15- monocytic MDSCs; Change at Week 4 | -0.1061 (0.22023)
  Myeloid-Derived Suppressor Cells (MDSC) panel: CD14+CD15- monocytic MDSCs; Change at Week 12: number analyzed (Participants) | 10
  Myeloid-Derived Suppressor Cells (MDSC) panel: CD14+CD15- monocytic MDSCs; Change at Week 12 | -0.1005 (0.25830)
  Myeloid-Derived Suppressor Cells (MDSC) panel: CD14+CD15- monocytic MDSCs; Change at Week 48: number analyzed (Participants) | 3
  Myeloid-Derived Suppressor Cells (MDSC) panel: CD14+CD15- monocytic MDSCs; Change at Week 48 | -0.3650 (0.41030)
  MDSC panel: CD124+ monocytic MDSCs; Baseline: number analyzed (Participants) | 10
  MDSC panel: CD124+ monocytic MDSCs; Baseline | 0.1525 (0.10414)
  MDSC panel: CD124+ monocytic MDSCs; Change at Week 4: number analyzed (Participants) | 5
  MDSC panel: CD124+ monocytic MDSCs; Change at Week 4 | -0.0536 (0.09398)
  MDSC panel: CD124+ monocytic MDSCs; Change at Week 12: number analyzed (Participants) | 6
  MDSC panel: CD124+ monocytic MDSCs; Change at Week 12 | -0.0816 (0.18479)
  MDSC panel: CD124+ monocytic MDSCs; Change at Week 48: number analyzed (Participants) | 2
  MDSC panel: CD124+ monocytic MDSCs; Change at Week 48 | -0.1308 (0.03511)
  MDSC panel: CD14-CD15+ granulocytic MDSCs; Baseline: number analyzed (Participants) | 10
  MDSC panel: CD14-CD15+ granulocytic MDSCs; Baseline | 0.3258 (0.36484)
  MDSC panel: CD14-CD15+ granulocytic MDSCs; Change at Week 4: number analyzed (Participants) | 9
  MDSC panel: CD14-CD15+ granulocytic MDSCs; Change at Week 4 | -0.0775 (0.30306)
  MDSC panel: CD14-CD15+ granulocytic MDSCs; Change at Week 12: number analyzed (Participants) | 8
  MDSC panel: CD14-CD15+ granulocytic MDSCs; Change at Week 12 | -0.1336 (0.45262)
  MDSC panel: CD14-CD15+ granulocytic MDSCs; Change at Week 48: number analyzed (Participants) | 5
  MDSC panel: CD14-CD15+ granulocytic MDSCs; Change at Week 48 | -0.0556 (0.34335)
  MDSC panel: CD124+ granulocytic MDSCs; Baseline: number analyzed (Participants) | 9
  MDSC panel: CD124+ granulocytic MDSCs; Baseline | 0.1689 (0.27247)
  MDSC panel: CD124+ granulocytic MDSCs; Change at Week 4: number analyzed (Participants) | 5
  MDSC panel: CD124+ granulocytic MDSCs; Change at Week 4 | -0.1310 (0.33046)
  MDSC panel: CD124+ granulocytic MDSCs; Change at Week 12: number analyzed (Participants) | 4
  MDSC panel: CD124+ granulocytic MDSCs; Change at Week 12 | -0.2081 (0.39793)
  MDSC panel: CD124+ granulocytic MDSCs; Change at Week 48: number analyzed (Participants) | 1
  MDSC panel: CD124+ granulocytic MDSCs; Change at Week 48 | 0.0380 (NA) — SD was not estimable as there was only one participant.
  MDSC panel: CD14-CD15- immature MDSCs; Baseline: number analyzed (Participants) | 9
  MDSC panel: CD14-CD15- immature MDSCs; Baseline | 0.2442 (0.20666)
  MDSC panel: CD14-CD15- immature MDSCs; Change at Week 4: number analyzed (Participants) | 7
  MDSC panel: CD14-CD15- immature MDSCs; Change at Week 4 | -0.0161 (0.21032)
  MDSC panel: CD14-CD15- immature MDSCs; Change at Week 12: number analyzed (Participants) | 4
  MDSC panel: CD14-CD15- immature MDSCs; Change at Week 12 | -0.1297 (0.18064)
  MDSC panel: CD14-CD15- immature MDSCs; Change at Week 48: number analyzed (Participants) | 5
  MDSC panel: CD14-CD15- immature MDSCs; Change at Week 48 | -0.0768 (0.13691)
  MDSC panel: CD124+ immature MDSCs; Baseline: number analyzed (Participants) | 4
  MDSC panel: CD124+ immature MDSCs; Baseline | 0.1011 (0.06344)
  MDSC panel: CD124+ immature MDSCs; Change at Week 4: number analyzed (Participants) | 2
  MDSC panel: CD124+ immature MDSCs; Change at Week 4 | -0.0853 (0.02369)
  Monocyte panel: CD14+CD16+; Baseline | 0.4317 (0.37154)
  Monocyte panel: CD14+CD16+; Change at Week 4: number analyzed (Participants) | 11
  Monocyte panel: CD14+CD16+; Change at Week 4 | -0.2408 (0.28990)
  Monocyte panel: CD14+CD16+; Change at Week 12: number analyzed (Participants) | 11
  Monocyte panel: CD14+CD16+; Change at Week 12 | -0.2424 (0.27183)
  Monocyte panel: CD14+CD16+; Change at Week 48: number analyzed (Participants) | 6
  Monocyte panel: CD14+CD16+; Change at Week 48 | 0.0250 (0.37069)
  Monocyte panel: CD14+CD16-; Baseline | 4.3404 (1.60025)
  Monocyte panel: CD14+CD16-; Change at Week 4 | -1.6758 (1.55056)
  Monocyte panel: CD14+CD16-; Change at Week 12: number analyzed (Participants) | 11
  Monocyte panel: CD14+CD16-; Change at Week 12 | -1.1205 (2.29278)
  Monocyte panel: CD14+CD16-; Change at Week 48: number analyzed (Participants) | 6
  Monocyte panel: CD14+CD16-; Change at Week 48 | -0.7592 (2.10992)
  Monocyte panel: CD14+HLA-DR+ CD11b+; Baseline | 4.5567 (1.62497)
  Monocyte panel: CD14+HLA-DR+ CD11b+; Change at Week 4 | -1.6504 (1.56493)
  Monocyte panel: CD14+HLA-DR+ CD11b+; Change at Week 12: number analyzed (Participants) | 11
  Monocyte panel: CD14+HLA-DR+ CD11b+; Change at Week 12 | -1.1155 (2.31024)
  Monocyte panel: CD14+HLA-DR+ CD11b+; Change at Week 48: number analyzed (Participants) | 6
  Monocyte panel: CD14+HLA-DR+ CD11b+; Change at Week 48 | -0.5925 (2.11151)
  Monocyte panel: CD14+HLA-DR+ CD163+; Baseline | 4.4613 (1.59602)
  Monocyte panel: CD14+HLA-DR+ CD163+; Change at Week 4 | -1.6679 (1.64311)
  Monocyte panel: CD14+HLA-DR+ CD163+; Change at Week 12: number analyzed (Participants) | 11
  Monocyte panel: CD14+HLA-DR+ CD163+; Change at Week 12 | -1.1223 (2.36705)
  Monocyte panel: CD14+HLA-DR+ CD163+; Change at Week 48: number analyzed (Participants) | 6
  Monocyte panel: CD14+HLA-DR+ CD163+; Change at Week 48 | -0.5167 (2.18389)
  Monocyte panel: CD14+HLA-DR+ CX3CR1+; Baseline | 4.3533 (1.54303)
  Monocyte panel: CD14+HLA-DR+ CX3CR1+; Change at Week 4 | -1.5529 (1.41647)
  Monocyte panel: CD14+HLA-DR+ CX3CR1+; Change at Week 12: number analyzed (Participants) | 11
  Monocyte panel: CD14+HLA-DR+ CX3CR1+; Change at Week 12 | -1.2809 (2.22435)
  Monocyte panel: CD14+HLA-DR+ CX3CR1+; Change at Week 48: number analyzed (Participants) | 6
  Monocyte panel: CD14+HLA-DR+ CX3CR1+; Change at Week 48 | -0.5992 (2.04927)

16. Secondary Outcome: Change From Baseline in Plasma Neurofilament Levels
Description: Levels of neurofilaments: Phosphorylated Neurofilament heavy chain (pNF-H) and Neurofilament light chain (NF-L) were measured by Enzyme-Linked Immunosorbent Assay (ELISA).
Time Frame: Baseline (Week 0), before and after PE procedure at Weeks 4, 12, 24, and before PE for Weeks 36 and 48
Population: Evaluable Population included all participants who received at least one PE treatment with albutein 5% and also had at least one baseline determination and measurement of a primary efficacy variable at a subsequent visit. Number analyzed is the number of participants with data available for analyses of the specific category at the given time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Albutein 5%
Number analyzed (Participants) | 12
ng/mL
  pNF-heavy, Baseline | 7.26 (5.811)
  pNF-heavy, Before PE Change at Week 4 | -1.29 (4.362)
  pNF-heavy, After PE Change at Week 4 | -5.46 (4.792)
  pNF-heavy, Before PE Change at Week 12: number analyzed (Participants) | 10
  pNF-heavy, Before PE Change at Week 12 | -0.99 (4.709)
  pNF-heavy, After PE Change at Week 12: number analyzed (Participants) | 10
  pNF-heavy, After PE Change at Week 12 | -4.97 (4.000)
  pNF-heavy, Before PE Change at Week 24: number analyzed (Participants) | 7
  pNF-heavy, Before PE Change at Week 24 | -0.93 (0.883)
  pNF-heavy, After PE Change at Week 24: number analyzed (Participants) | 7
  pNF-heavy, After PE Change at Week 24 | -3.39 (2.265)
  pNF-heavy, Before PE Change at Week 36: number analyzed (Participants) | 8
  pNF-heavy, Before PE Change at Week 36 | 0.47 (3.526)
  pNF-heavy, Before PE Change at Week 48: number analyzed (Participants) | 6
  pNF-heavy, Before PE Change at Week 48 | 1.50 (2.471)
  NF-light, Baseline | NA (NA) — Data is not available as NF-light concentration levels were below the level of detection.
  NF-light, Before PE Change at Week 4 | NA (NA) — Data is not available as NF-light concentration levels were below the level of detection.
  NF-light, After PE Change at Week 4 | NA (NA) — Data is not available as NF-light concentration levels were below the level of detection.
  NF-light, Before PE Change at Week 12: number analyzed (Participants) | 10
  NF-light, Before PE Change at Week 12 | NA (NA) — Data is not available as NF-light concentration levels were below the level of detection.
  NF-light, After PE Change at Week 12: number analyzed (Participants) | 10
  NF-light, After PE Change at Week 12 | NA (NA) — Data is not available as NF-light concentration levels were below the level of detection.
  NF-light, Before PE Change at Week 24: number analyzed (Participants) | 7
  NF-light, Before PE Change at Week 24 | NA (NA) — Data is not available as NF-light concentration levels were below the level of detection.
  NF-light, After PE Change at Week 24: number analyzed (Participants) | 7
  NF-light, After PE Change at Week 24 | NA (NA) — Data is not available as NF-light concentration levels were below the level of detection.
  NF-light, Before PE Change at Week 36: number analyzed (Participants) | 8
  NF-light, Before PE Change at Week 36 | NA (NA) — Data is not available as NF-light concentration levels were below the level of detection.
  NF-light, Before PE Change at Week 48: number analyzed (Participants) | 6
  NF-light, Before PE Change at Week 48 | NA (NA) — Data is not available as NF-light concentration levels were below the level of detection.

17. Secondary Outcome: Change From Baseline in Cerebrospinal Fluid (CSF) Neurofilament Levels
Description: as for outcome 16
Time Frame: Baseline (Week 0), Weeks 12, and 25
Population: Evaluable Population included all participants who received at least one PE treatment with albutein 5% and also had at least one baseline determination and a measurement of a primary efficacy variable at a subsequent visit. Number analyzed is the number of participants with data available for analyses for the specific category at the given time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Albutein 5%
Number analyzed (Participants) | 12
ng/mL
  pNF-heavy, Baseline | 0.68 (0.147)
  pNF-heavy, Change at Week 12: number analyzed (Participants) | 11
  pNF-heavy, Change at Week 12 | -0.01 (0.130)
  pNF-heavy, Change at Week 25: number analyzed (Participants) | 7
  pNF-heavy, Change at Week 25 | 0.07 (0.160)
  NF-light, Baseline | 7463.0 (5857.49)
  NF-light, Change at Week 12: number analyzed (Participants) | 11
  NF-light, Change at Week 12 | 270.6 (496.12)
  NF-light, Change at Week 25: number analyzed (Participants) | 7
  NF-light, Change at Week 25 | 823.0 (1137.62)

18. Other Pre Specified Outcome: Percentage of PE Sessions Associated With at Least One Adverse Reaction (AR)
Time Frame: During or within 72 hours after the completion of the product infusion
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Percentage of PE Sessions Associated With at Least One Adverse Event (AE), Irrespective of Causality
Time Frame: During or within 72 hours after the completion of the product infusion
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Incidence of All AEs
Time Frame: Weeks -2 to 48
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the start of study treatment until end of study (Up to Week 48)
Description: Safety population included all participants who received any amount of the study drug.
Arm/Group | Albutein 5%
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albutein 5% (N=12)
Jugular vein occlusion (Nervous system disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albutein 5% (N=12)
Conjunctival haemorrhage (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Inguinal hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Retching (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Catheter site erythema (General disorders) | 1
Catheter site inflammation (General disorders) | 1
Catheter site pain (General disorders) | 1
Catheter site pruritus (General disorders) | 1
Catheter site related reaction (General disorders) | 1
Chest discomfort (General disorders) | 1
Fatigue (General disorders) | 2
Feeling hot (General disorders) | 1
Gait disturbance (General disorders) | 2
Oedema peripheral (General disorders) | 3
Peripheral swelling (General disorders) | 2
Concussion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 4
Head injury (Injury, poisoning and procedural complications) | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 3
Skin laceration (Injury, poisoning and procedural complications) | 2
Wound complication (Injury, poisoning and procedural complications) | 1
Blood calcium decreased (Investigations) | 2
Blood fibrinogen decreased (Investigations) | 2
Blood potassium decreased (Investigations) | 2
Weight decreased (Investigations) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Masticatory pain (Musculoskeletal and connective tissue disorders) | 1
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Balance disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 5
Dysarthria (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Muscle contractions involuntary (Nervous system disorders) | 1
Muscular weakness (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Cold sweat (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Livedo reticularis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Scab (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 2
Venous thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2016-05-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT02872142/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT02872142/SAP_001.pdf